CLINICAL TRIAL: NCT07016425
Title: Efficacy and Safety of Non-invasive Temporal Interference Stimulation in the Treatment of Essential Tremor: A Pilot Trial
Brief Title: Temporal Interference for Essential Tremor
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Liankun_Ren (Other)
Responsible Party: Sponsor-Investigator, Liankun_Ren, Professor, Xuanwu Hospital, Beijing
Organization: Xuanwu Hospital, Beijing (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-426-002
Record Dates: First submitted 2025-06-03; First posted 2025-06-11 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Essential Tremor
Keywords: Temporal Interference; Essential Tremor
MeSH Terms: conditions — Essential Tremor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Temporal Interference (Experimental): The investigators perform temporal interference (TI) stimulation to patients with essential tremor. They observe clinical manifestations before and after stimulation to investigate the efficiency of TI.
  Interventions: Other: Temporal Interference

INTERVENTIONS:
Other: Temporal Interference — Researchers apply temporal interference (TI) stimulation to the deep brain nuclei of essential tremor patients.

SUMMARY:
This single-center prospective study aims to investigate the treatment efficacy of temporal interference (TI) in essential tremor patients aged 30-70.

DETAILED DESCRIPTION:
Temporal Interference (TI) technology is a novel non-invasive method for deep brain stimulation (DBS). By generating an overlapping electric field from safe currents, TI creates focused stimulation in targeted deep brain areas. This approach allows for the exploration of deep brain nuclei functions and has the potential to serve as a non-invasive alternative to traditional invasive DBS for clinical treatments.

This study aims to investigate the treatment efficacy of TI deep brain stimulation by including essential tremor patients aged 30-70. Before and after TI stimulation, clinical data will be recorded. Clinical and imaging data will be analyzed and processed to advance the treatment of essential tremor.

ELIGIBILITY:
Inclusion Criteria:

* Aged 30-70 years old, regardless of gender. Action tremor and postural tremor in both upper limbs, or action tremor and postural tremor in one limb;
* No history of mental diseases;
* Informed consent signed.

Exclusion Criteria:

* Presence of other neurological diseases affecting the study (such as epilepsy);
* Patients with moderate to severe cognitive impairment (Montreal Cognitive Assessment ≤ 18 points);
* Orthopedic diseases that may affect motor symptoms;
* Patients taking antipsychotic or antidepressant medications;
* Presence of metal implants in the body (such as brain pacemakers or cardiac pacemakers);
* History of electroconvulsive therapy;
* Presence of cardiovascular risk factors, etc.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-06-09 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Tremor Level Evaluation | Up to 3 months after TI stimulation
  Percentage change in per month after stimulation from baseline in The Essential Tremor Rating Assessment Scale(TETRAS) score. The TETRAS score ranges from 0 to 112, including an activities of daily living (ADL) section(0-48 scores) and a performance section(0-64 scores), with higher scores representing more severe tremor and lower scores indicating lower tremor level

CONTACTS AND LOCATIONS:
Overall Officials: Liankun Ren, MD, Principal Investigator — Xuanwu Hospital, Beijing
Locations (1):
- Xuanwu Hospital, Capital Medical University, Beijing, Beijing Municipality, China